CLINICAL TRIAL: NCT00241163
Title: An Open, Randomised, Prospective, Multicentre, Parallel-group Trial to Compare Efficacy and Safety of TachoComb S Versus Standard Surgical Treatment in Patients Undergoing Surgical Resection of Superficial Renal Tumour.
Brief Title: TachoComb S Versus Standard Surgical Treatment in Surgical Resection of Renal Tumour (TC-015-IN)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TC-015-IN
Record Dates: First submitted 2005-10-16; First posted 2005-10-18 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-05

CONDITIONS: Surgical Resection of Superficial Renal Tumour
MeSH Terms: interventions — Fibrinogen; Thrombin; TachoSil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Fibrinogen (human) + thrombin (human) (TachoSil)

SUMMARY:
The overall objective is to compare efficacy and safety of TachoComb S and standard surgical treatment for the control of local bleeding in patients undergoing surgical resection of renal tumours. Specific objectives include the comparison between test treatments of intra-operative haemostatic efficacy as well as post-operative blood loss, haematoma formation, and surgeon's rating of usefulness of test treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients of or above 18 years of age scheduled for resection of superficial tumour on the kidney and scheduled for open surgery. After the tumour resection the wound should be suitable for the treatments in the study, and the integrity of the urinary tract should be maintained.

Exclusion criteria:

Patients undergoing an emergency operation, or with more than one tumour will be excluded. Patients with a clinically abnormal value of prothrombin time or activated partial thromboplastin time, anamnetic evidence of coagulation disorders and a history of allergic reactions after application of human fibrinogen, human thrombin and/or collagen will be excluded. In case the tumour was resected by use of a laser scalpel, infrared coagulator or argon beamer and if any fibrin glue haemostatic was used before randomisation the patient will be excluded from the trial. Furthermore, patients will be excluded if extensive resection/extirpation of the kidney become necessary or in case of serious surgical complication occurring during the operation.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170

PRIMARY OUTCOMES:
Primary efficacy endpoint is overall time to intraoperative haemostasis from start of test treatment until haemostasis is obtained following 1 or 2 rounds of randomised treatment,and other haemostatic treatment, if necessary.

SECONDARY OUTCOMES:
Secondary efficacy endpoints are: 1) proportion of patients with haemostasis 10 minutes after start of test treatment; 2) haematoma formation on day 2 after surgery (sonography).
Adverse events will be recorded from screening until follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Please refer to this study by ClinicalTrials.gov identifier NCT00241163, Nycomed, Study Chair — Takeda
Locations (1):
- Roskilde, Denmark